CLINICAL TRIAL: NCT04020263
Title: Effect of Early Use of Levosimendan Versus Placebo on Top of a Conventional Strategy of Inotrope Use on a Combined Morbidity-mortality Endpoint in Patients With Cardiogenic Shock
Acronym: LevoHeartShock
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pr Bruno LEVY (Other)
Responsible Party: Sponsor-Investigator, Pr Bruno LEVY, Investigator coordonnator, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-513811-29-00; 2024-513811-29-00 (EU CTIS Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cardiogenic Shock
Keywords: heart failure; levosimendan
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure | interventions — Simendan

STUDY DESIGN:
Intervention Model Description: The LevoHeartShock trial is a prospective, double-blind, multicenter, randomized controlled trial comparing the early initiation of levosimendan versus placebo in patients with cardiogenic shock treated with vasopressor therapy according to a conventional strategy of inotrope use (dobutamine as first line agent).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be double-blinded. Investigator masking to group assignment after randomization will be guaranteed by use of a placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimendan (Experimental): Experimental group: patients with cardiogenic shock treated with levosimendan in addition to the conventional strategy.
  Interventions: Drug: Levosimendan 2.5 MG/ML Injectable Solution
- Placebo (Placebo Comparator): Control group: Patients with cardiogenic shock treated with placebo (Cernevit/Soluvit) in addition to the conventional strategy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan 2.5 MG/ML Injectable Solution — Levosimendan will be diluted with Glucose G5%. The reconstitution of levosimendan will be performed, as close as possible to the start of the infusion. A continuous infusion of levosimendan will be administered over 24 h without bolus, started at a rate of 0.1 μg per kilogram of body weight per minute and, in both the persistence of hypoperfusion signs and in the absence of rate-limiting side effects, will be increased after 2 to 4 hours to a maximum of 0.2 μg per kilogram per minute for a further 20 to 22 hours.
  Arms: Levosimendan
Drug: Placebo — Placebo will be diluted with Glucose G5%. The reconstitution of Placebo will be performed, as close as possible to the start of the infusion. A continuous infusion of Placebo will be administered over 24 h without bolus, started at a rate of 0.1 μg per kilogram of body weight per minute and, in both the persistence of hypoperfusion signs and in the absence of rate-limiting side effects, will be increased after 2 to 4 hours to a maximum of 0.2 μg per kilogram per minute for a further 20 to 22 hours.
  Arms: Placebo

SUMMARY:
Cardiogenic shock (CS) mortality remains high (40%). Despite their frequent use, few clinical outcome data are available to guide the initial selection of vasoactive drug therapies in patients with CS. Based on experts' opinions, the combination of norepinephrine-dobutamine is generally recommended as a first line strategy. Inotropic agents increase myocardial contractility, thereby increasing cardiac output. Dobutamine is commonly recommended to be the inotropic agent of choice and levosimendan is generally used following dobutamine failure. It may represent an ideal agent in cardiogenic shock, since it improves myocardial contractility without increasing cAMP or calcium concentration. At present, there are no convincing data to support a specific inotropic agent in patients with cardiogenic shock. Our hypothesis is that the early use of levosimendan, by enabling the discontinuation of dobutamine, would accelerate the resolution of signs of low cardiac output and facilitate myocardial recovery.

ELIGIBILITY:
Inclusion Criteria:

Adult patient ≥ 18 years with cardiogenic shock defined by:

* Adequate intravascular volume
* Norepinephrine to maintain MAP at least at 65 mmHg for at least 3 hours and less than 24h. At inclusion the dose must be <1 microgram/kg/min under norepinephrine base or <2 microgram/kg/min under norepinephrine tartrate, OR/AND Dobutamine since at least 3h and less than 24h at inclusion.
* Tissue hypoperfusion: at least 1 sign within 24h prior to inclusion (lactate ≥ 2 mmol/l; mottling, capillary refeel time > 3 seconds, oliguria <500ml/24h or ≤ 20 ml/h during the last 2 hours, ScVO2 ≤ 60% or veno-arterial PCO2 gap ≥ 5 mmHg);

Exclusion Criteria:

* Myocardial sideration after cardiac arrest of non-cardiac etiology
* Immediate or anticipated (within 6 hours) indication of Extra Corporel Life Support
* Use of VA-ECMO or IMPELLA or LVAD;
* Chronic renal failure requiring hemodialysis
* Cardiotoxic poisoning
* Septic cardiomyopathy
* Previous levosimendan administration within 15 days
* Cardiac arrest with non-shockable rhythm;
* No flow time higher > 3 minutes;
* Cardiac arrest with unknown no flow duration;
* Total duration of cardiac arrest (no flow plus low flow) > 45 minutes;
* Cerebral deficit with fixed dilated pupils
* Patient moribund on the day of enrollment
* Irreversible neurological pathology
* Known hypersensitivity to levosimendan or placebo, or one of its excipients
* Pregnant woman, birthing or breastfeeding mother
* Minor (not emancipated)
* Person deprived of liberty for judicial or administrative decision;
* Adult subject to a legal protection measure (such as guardianship, conservatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-02-03 (Estimated); Study Completion 2028-01-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of All-cause mortality | Day 30 following randomization
  Composite endpoint (i.e. All-cause Mortality and/or Extra Corporel Life Support implantation and/or dialysis)
Proportion of Extra Corporel Life Support implantation | Day 30 following randomization
  Composite endpoint (i.e. All-cause Mortality and/or Extra Corporel Life Support implantation and/or dialysis)
Proportion of Dialysis | Day 30 following randomization
  Composite endpoint (i.e. All-cause Mortality and/or Extra Corporel Life Support implantation and/or dialysis)

SECONDARY OUTCOMES:
Time to death | Day 90
  Prioritized composite endpoint with the following priority order: 1/ time to death, 2/ escalation to permanent left ventricular assist device or cardiac transplantation, 3/ dialysis, 4/ ECLS requirement, 5/ number of cardiovascular events (stroke, recurrent myocardial infarction, urgent coronary revascularization, re-hospitalization for heart failure).
Time to escalation to permanent left ventricular assist device or cardiac transplantation | Day 90
  Prioritized composite endpoint with the following priority order: 1/ time to death, 2/ escalation to permanent left ventricular assist device or cardiac transplantation, 3/ dialysis, 4/ ECLS requirement, 5/ number of cardiovascular events (stroke, recurrent myocardial infarction, urgent coronary revascularization, re-hospitalization for heart failure).
Time to dialysis | Day 90
  Prioritized composite endpoint with the following priority order: 1/ time to death, 2/ escalation to permanent left ventricular assist device or cardiac transplantation, 3/ dialysis, 4/ ECLS requirement, 5/ number of cardiovascular events (stroke, recurrent myocardial infarction, urgent coronary revascularization, re-hospitalization for heart failure).
Time to ECLS requirement | Day 90
  Prioritized composite endpoint with the following priority order: 1/ time to death, 2/ escalation to permanent left ventricular assist device or cardiac transplantation, 3/ dialysis, 4/ ECLS requirement, 5/ number of cardiovascular events (stroke, recurrent myocardial infarction, urgent coronary revascularization, re-hospitalization for heart failure).
number of cardiovascular events | Day 90
  Prioritized composite endpoint with the following priority order: 1/ time to death, 2/ escalation to permanent left ventricular assist device or cardiac transplantation, 3/ dialysis, 4/ ECLS requirement, 5/ number of cardiovascular events (stroke, recurrent myocardial infarction, urgent coronary revascularization, re-hospitalization for heart failure).
Proportion of death. | Day 90
Proportion of Extra Corporel Life Support implantation | Day 90
Proportion of dialysis | Day 90
Proportion of cardiac transplantation | Day 90
Proportion of escalation to permanent Left Ventricular Assist Device | Day 90
Proportion of stroke | Day 90
Proportion of recurrent myocardial infarction | Day 90
Proportion of urgent coronary revascularization | Day 90
Proportion of re-hospitalization for heart failure | Day 90
Proportion of All-cause mortality | Day 90
  Composite endpoint of all-cause mortality and/or ECLS requirement and/or dialysis on day 90.
Proportion of Extra Corporel Life Support implantation | Day 90
  Composite endpoint of all-cause mortality and/or ECLS requirement and/or dialysis on day 90.
Proportion of Dialysis | Day 90
  Composite endpoint of all-cause mortality and/or ECLS requirement and/or dialysis on day 90.
Number of dobutamine free days | From randomization to day 30
Number of vasopressors free days | From randomization to day 30
Number of ventilatory free days | From randomization to day 30
Number of renal replacement free days | From randomization to day 90
Lactate clearance | from randomization to day 7
Duration of intensive care unit stay | Up to Intensive Care Unit discharge (assessed up to 1 month)
Duration of hospitalization | Up to hospitalization discharge (assessed up to 1 month)
Proportion of All-cause mortality | days 7, 60, and 180 days and 12 months
  Composite endpoint of all-cause mortality and/or ECLS requirement and/or dialysis
Proportion of Extra Corporel Life Support implantation | days 7, 60, and 180 days and 12 months
  Composite endpoint of all-cause mortality and/or ECLS requirement and/or dialysis
Proportion of dialysis | days 7, 60, and 180 days and 12 months
  Composite endpoint of all-cause mortality and/or ECLS requirement and/or dialysis
Number of renal replacement free days | D 30, 60, 180 and at 12 months
Proportion of death | days 180 and at 12 months
Proportion of Extra Corporel Life Support implantation | days 180 and at 12 months
Proportion of dialysis | days 180 and at 12 months
proportion of cardiac transplantation | days 180 and at 12 months
proportion of escalation to permanent left ventricular assist device | days 180 and at 12 months
Proportion of stroke | days 180 and at 12 months
Proportion of recurrent myocardial infarction | days 180 and at 12 months
Proportion urgent coronary revascularization | days 180 and at 12 months
proportion of re-hospitalization for heart failure | days 180 and at 12 months
Occurrence of arrhythmias requiring therapy | from randomization to intensive care unit discharge.
  Occurrence of arrhythmias requiring therapy with anti-arrhythmic drugs or electric cardioversion (including atrial fibrillation, ventricular tachycardia, ventricular fibrillation, torsade de pointe)
the changes in biomarkers | from randomization to intensive care unit discharge.
  From a dedicated biological collection on which we will measure existing and future biological parameters, we will evaluate the effect of Levosimendan on the changes in biomarkers between randomization and ICU/CCU discharge
All-cause mortality and/or ECLS and/or dialysis | Day 30
  From a dedicated biological collection on which we will measure existing and future biological parameters, we will evaluate the ability of clinical and biological measure to predict levosimendan effect for the primary endpoint.
All-cause mortality and/or ECLS and/or dialysis | At intensive care unit discharge
  From a dedicated biological collection on which we will measure existing and future biological parameters, we will evaluate the ability of biological measure to predict subsequent outcome

CONTACTS AND LOCATIONS:
Overall Officials: Clément DELMAS, Dr, Study Chair — University Hospital, Toulouse; Nicolas GIRERD, Pr, Study Chair — CHRU Nancy; Patrick ROSSIGNOL, Pr, Study Chair — CHRU Nancy
Locations (28):
- France (28):
  - CHRU Strasbourg -Nouvel Hôpital Civil, Strasbourg, Bas-Rhin
  - AP-HM, Nord Hospital, Marseille, Marseille, Bouches du Rhône
  - CHU Caen, Caen, Calvados
  - CHU Dijon, Dijon, Côte d'Or
  - CHU Besançon Jean Minjoz Hospital, Besançon, Doubs
  - CHU Nîmes, Carémeau Hospital, Nîmes, Gard
  - CHU Bordeaux - Hopital haut-leveque, Bordeaux, Gironde
  - CHU de Toulouse, Toulouse, Haute-Garonne
  - CHU Limoges, Dupuytren Hospital, Limoges, Haute-Vienne
  - CHU Montpellier, Arnaud de Villeneuve Hospital, Montpellier, Hérault
  - CHU Rennes, Pontchaillou Hospital, Rennes, Ille et Vilaine
  - CHU Grenoble, Michallon Hospital, La Tronche, Isère
  - CHU Nantes, Nantes, Loire-Atlantique
  - CHR Metz-Thionville, Mercy Hospital, Ars-Laquenexy, Moselle
  - CHRU Lille, Cœur Poumon Institute, Lille, Nord
  - APHP, La Pitié Salpêtrière (medical intensive care unit), Paris, Paris
  - Hospices Civils de Lyon - Louis Pradel Hospital, Bron, Rhône
  - APHP, Henri Mondor Hospital, Créteil, Val de Marne
  - CH Henri Duffaut, Avignon, Avignon, Vaucluse
  - CHU Bordeaux, Bordeaux
  - HENRI MONDOR -réanimation, Créteil
  - Chu Dijon, Dijon
  - CHU Grenoble -USIC, La Tronche
  - AP-HM CHU la Timone, Marseille
  - CHU Montpellier -hôpital Arnaud de Villeneuve, Montpellier
  - Chu Rouen, Rouen
  - HU Strasbourg USIC, Strasbourg
  - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided